CLINICAL TRIAL: NCT01551316
Title: A Phase Ib Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of Repeated Administration, Intravenous MN-221 in Stable Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Safety Study to Evaluate MN-221 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MN-221-CL-012
Record Dates: First submitted 2012-02-08; First posted 2012-03-12 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: safety; pharmacokinetics; spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — bedoradrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MN-221 (Experimental): If the participants qualify, they will be randomized into one of two arms for 4 days. The arms are either Placebo (no medication) or MN-221 intravenously infused.
  Interventions: Drug: MN-221
- PLACEBO (Experimental): If the participants qualify, they will be randomized into one of two arms for 4 days. The arms are either Placebo (no medication) or MN-221 intravenously infused.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MN-221 — This drug is intravenously infused and delivers 1200 mcg to the patient in 1 hour duration. This dose is repeated over 4 days (Day 1 1200 mcg once; Day 2 1200 mcg twice; Day 3 1200 mcg twice; Day 4 1200 mcg once).
  Other Names: Bedoradrine Sulfate
  Arms: MN-221
Drug: Placebo — This intervention consists of a placebo intravenous infusion, one that contains no active medication. During the double-blind procedure, patients will be infused with placebo intravenously one time on Day 1, twice on Days 2 and 3, and one time on Day 4.
  Arms: PLACEBO

SUMMARY:
In MediciNova's clinical development plan for MN-221, it was recognized that treatment of COPD exacerbations may necessitate more than one single i.v. infusion and that patients in this population may have more co-morbidities (and concomitant medications) than has been generally studied so far. Thus, the primary objective of this clinical study is to determine the repeated administration safety and tolerability of intravenous (i.v.) MN-221 compared to placebo with repeated administration over several days in moderate to severe COPD patients who may also have co-morbidities and concomitant medications (CM) common in this population. Secondary outcomes include pharmacokinetics (PK) and preliminary efficacy (FEV1).

This Phase 1b trial follows naturally upon a Phase 1b COPD trial completed last year (MN-221-CL-010) and is additionally well-supported by relevant animal safety data and human clinical trial information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 40-75 years of age, inclusive;
* History of physician-diagnosed (e.g., by clinical history, >15-pack year history of smoking, physical examination, and spirometry) COPD treated for ≥ 3 months prior to Visit 1 Pre-Screening;
* FEV1 ≥ 30% and < 80% predicted and FEV1/FVC ratio < 0.7 at Visit 1 Pre-Screening and Visit 2 Screening;
* Negative urine pregnancy test for all females unless the subject is post-menopausal (≥ 24 months of spontaneous amenorrhea) or surgically sterile (hysterectomy, bilateral ovariectomy or bilateral tubal ligation);
* Negative urine drug screen for cocaine, phencyclidine (PCP), methamphetamine;
* Negative alcohol breath test;
* Electrocardiogram (ECG) without serious abnormality and with QTcB and QTcF < 460 milliseconds (msec);
* Ability to wash-out of concomitant LABA and Theophylline, if ongoing, for 7-8 days (i.e., Visit 2 Screening through 5-Day Treatment Period).
* Legally effective written informed consent obtained prior to starting any study procedures.
* Subject willing and able to comply with the protocol and procedures, as judged by Investigator.

Exclusion Criteria:

* Sustained release methylxanthine (e.g. Theophylline) or long acting beta agonists ≤ 48 hours prior to treatment start (Day 1);
* Acute exacerbation of COPD requiring emergency treatment ≤ 30 days of screening or hospitalization ≤ 60 days of Visit 2 Screening;
* Antibiotic therapy for respiratory infection ≤ 15 days of Visit 2 Screening;
* Presence of active respiratory disease such as pneumonia and acute exacerbation of chronic bronchitis;
* Hypokalemia defined as a potassium level <3.0 mmol/L at Visit 2 Screening. note: Subjects <3.0 mmol/L may be re-screened at Visit 2 Screening after receiving potassium replacement therapy;
* Significant clinical laboratory abnormality that, in the opinion of the Investigator, may put the subject at risk;
* Significant renal, hepatic, endocrine, neurologic or other systemic disease that, in the opinion of the Investigator, may put the subject at undue risk;
* Uncontrolled hypertension (defined as a blood pressure ≥ 170/100 mm Hg at Visit 1 Pre-Screening) and/or uncontrolled angina, uncontrolled diabetes, uncontrolled congestive heart failure (CHF), uncontrolled serious arrhythmia;
* Myocardial infarction within 6 months of treatment start;
* Pregnant or lactating females;
* Participation in another clinical study with an investigational drug within 30 days of Visit 1 Pre-Screening;
* Patients with home oxygen requirements.
* A known allergy to excipients of the MN-221 drug product;
* A known allergy to other beta agonists;
* Currently on medication/s that are recognized to have risk of Torsades de Pointes

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Treatment Days 1- 5
  The recording of AEs will start after the subject has signed the consent form and will end at the Hour 24 phone interview. Investigator(s) will monitor each subject closely for AEs and the Investigator will record all observed or volunteered AEs.

SECONDARY OUTCOMES:
MN-221 and primary metabolite levels will be analyzed by liquid chromatography/mass spectrometry/mass spectrometry. | Treatment Days 1-5
  Blood samples will be analyzed for MN-221 and primary metabolite levels by liquid chromatography/mass spectrometry (LC/MS/MS.
Evaluation of respiratory parameters (FEV1, peak flow, accessory muscle use, respiratory rate) | Screening, Treatment Days 1,3,5

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas